CLINICAL TRIAL: NCT06904664
Title: Individualized Temperature Health Risk Early Warning and Risk Factor Management App for Reducing the Recurrence Risk of Stroke: A Multicenter, Randomized Controlled Trial Study
Brief Title: An Application That Can Provide Early Warning of Temperature Health Risks and Give Protective Suggestions or Personalized Suggestions Based on Patients' Own Secondary Prevention Risk Factors Was Applied to Intervene, and the Intervention Effect of APP on Stroke Recurrence Risk Was Analyzed
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: [2024]444-003-1-3
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced intervention group (Experimental): Receive individualized temperature health risk warning and prevention risk factor management information for stroke through the application
  Interventions: Other: Individualized temperature health risk early warning and risk factor management
- Temperature health risk early warning group (Experimental): Receive individualized temperature health risk warning through the application
  Interventions: Other: Temperature health risk early warning
- Risk factor management group (Experimental): Receive individualized prevention risk factor management information for stroke through the application
  Interventions: Other: Risk factor management
- Routine education group (No Intervention): Only receive routine health education, without receiving individualized temperature health risk warning or prevention risk factor management information for stroke through the application

INTERVENTIONS:
Other: Individualized temperature health risk early warning and risk factor management — Receive individualized temperature health risk warning and prevention risk factor management information for stroke through the application
  Arms: Enhanced intervention group
Other: Temperature health risk early warning — Receive individualized temperature health risk warning through the application
  Arms: Temperature health risk early warning group
Other: Risk factor management — Receive individualized prevention risk factor management information for stroke through the application
  Arms: Risk factor management group

SUMMARY:
This study employs individualized temperature health risk early warning and risk factor management interventions for stroke, and explores their actual intervention effects. This enables patients to promptly understand their own risk levels and take corresponding protective measures, thereby enhancing the management outcomes and quality of life. The study also promotes the interdisciplinary integration of environmental epidemiology and clinical intervention management, providing new ideas and methodological support for future relevant research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 80, with no gender restrictions;

  * Acute ischemic stroke inpatients within 2 weeks of onset, where the onset time is the time when stroke symptoms appear or the last known normal time of the patient (when it is an onset during sleep or the symptom onset time cannot be accurately obtained due to aphasia, impaired consciousness, etc.); ③ Confirmed diagnosis of ischemic stroke by CT or MRI of the brain within 2 weeks after symptom onset;

    * Local residents (residing for ≥6 months); ⑤ Patients who voluntarily participate in the study, have high compliance, and can sign the informed consent form;

      * Patients who own a smartphone or other smart devices.

Exclusion Criteria:

* Patients diagnosed with other cerebrovascular diseases (hemorrhagic stroke, transient ischemic attack, cerebral venous sinus thrombosis, etc.) or non-cerebrovascular diseases;

  * Known pregnant or lactating women, or those who tested positive on a pregnancy test before cluster randomization;

    * Patients with other conditions that may affect participation in the trial (e.g., refractory hypertension, severe aphasia, etc.);

      * Patients undergoing psychiatric/psychological treatment that may contaminate the results; ⑤ Patients with a life expectancy of less than one year (e.g., coexisting malignant tumors, severe cardiopulmonary diseases, etc.); ⑥ Patients already participating in other interventional clinical studies that may influence the outcome assessment; ⑦ Patients for whom the investigator deems unsuitable for participation in this study or who may pose significant risks to the patients (e.g., cognitive impairment preventing understanding and/or compliance with the study procedures and/or follow-up).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10184 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence rate of stroke | Intervention at the 1-year

SECONDARY OUTCOMES:
3-month, 6-month, 9-month recurrence rate of stroke | Intervention at 3-month, 6-month, 9-month
Cardiovascular system function indicators | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Such as blood pressure, various electrocardiogram indicators and other examination results that can reflect cardiovascular function
Laboratory examination | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Such as results of laboratory tests including lipid profiles, blood glucose, coagulation, and other laboratory indicators.
Modified Rankin Scale | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  The Modified Rankin Scale (mRS) is a scale used to assess the neurological recovery status and disability level in stroke patients. The scale ranges from zero to six, divided into seven levels, with higher grades indicating worse conditions.
European five-dimensional five-level Health Scale score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  The scale includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with each dimension containing five levels. It also includes a 0-100 scale, where a lower score indicates worse condition.
Risk perception scale of stroke recurrence | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  The scale uses a Likert three-point scoring method, assigning values of 1, 2, and 3 for the responses "disagree," "uncertain," and "agree," respectively. A higher score indicates a higher level of perceived ability.
Environmental temperature health risk perception assessment 1uestionnaire | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Here are multiple questions related to environmental risk factors and health risks, each using a 0-100 scale where a higher score indicates greater understanding
Stroke health literacy score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  The scale uses a five-point scoring method, with a higher score indicating a higher level of stroke health literacy.
Health status score | Baseline; Intervention at 3-month, 6-month, 9-month and 1-year
  Such as barthel index (BI) and other scoring scales for evaluating patients' disease recovery, physical condition and other abilities
System usability scale | Intervention at 3-month, 6-month, 9-month and 1-year

OTHER OUTCOMES:
Incidence of adverse cerebrovascular events | Intervention at the 1-year

IPD SHARING:
Plan to Share IPD: No